CLINICAL TRIAL: NCT01668966
Title: A Multicenter, Open-Label, Single Arm, Long Term Extension Study of WA19926 to Describe Safety During Treatment With Tocilizumab in Patients With Early, Moderate to Severe Rheumatoid Arthritis
Brief Title: A Long Term Extension Study of WA19926 (NCT01007435) of Tocilizumab (RoActemra/Actemra) in Participants With Early, Moderate to Severe Rheumatoid Arthritis (RA)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML28080
Record Dates: First submitted 2012-08-16; First posted 2012-08-20 (Estimated); Results first posted 2019-05-13 (Actual); Last update posted 2019-05-13 (Actual); Status verified 2019-02

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — tocilizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tocilizumab (Experimental): Participants will receive tocilizumab 8 milligrams per kilogram (mg/kg) intravenously (IV) every 4 weeks for up to 104 weeks.
  Interventions: Drug: Tocilizumab

INTERVENTIONS:
Drug: Tocilizumab — Participants will receive tocilizumab 8 mg/kg IV every 4 weeks for up to 104 weeks.
  Other Names: RoActemra, Actemra

SUMMARY:
This open-label, single arm, multicenter long-term extension study of WA19926 (NCT01007435) will evaluate the safety and efficacy of tocilizumab in participants with early, moderate to severe RA who have completed the 104-week WA19926 (NCT01007435) core study. Eligible participants will be those who are expected to benefit from the study medicine based on the investigator's discretion.

ELIGIBILITY:
Inclusion Criteria:

* Participants who completed their last WA19926 (NCT01649804) core study visit (Week 104) and who may benefit from study drug treatment according to the Investigator's assessment
* No current or recent adverse event or laboratory finding preventing the use of tocilizumab 8 mg/kg at baseline visit
* Women of childbearing potential must agree to use highly reliable contraception during the treatment period

Exclusion Criteria:

* Pregnant or breastfeeding females
* Participants who have withdrawn prematurely from the WA19926 (NCT01649804) core study for any reason
* Treatment with any investigational agent or cell-depleting therapies since the last administration of study drug in WA19926 (NCT01649804)
* Treatment with an anti-tumor necrosis factor (TNF) or anti-interleukin (IL) 1 agent, or a T-cell costimulation modulator since the last administration of study drug in WA19926 (NCT01649804)
* Immunization with a live/attenuated vaccine since the last administration of study drug in WA19926 (NCT01649804)
* Diagnosis since last WA19926 (NCT01649804) visit (Week 104) of rheumatic autoimmune disease other than RA
* Diagnosis since last WA19926 (NCT01649804) visit (Week 104) of inflammatory joint disease other than RA
* History of severe allergic or anaphylactic reactions to humanized or murine monoclonal antibodies, including tocilizumab and its excipients
* Evidence of severe uncontrolled concomitant disease or disorder
* Known active infections or history of recurrent infections
* Active tuberculosis requiring treatment in the previous 3 years
* History of alcohol, drug or chemical abuse since inclusion in the WA19926 (NCT01649804) study

Min Age: 18 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2013-12-09 (Actual); Primary Completion 2016-05-11 (Actual); Study Completion 2016-05-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (6):
- Brazil (6):
  - CIP - Centro Internacional de Pesquisa, Goiânia, Goiás
  - Centro Mineiro de Pesquisa - CMIP, Juiz de Fora, Minas Gerais
  - Centro de Estudos em Terapias Inovadoras - CETI, Curtiba, Paraná
  - Hospital Sao Lucas - PUCRS, Porto Alegre, Rio Grande do Sul
  - Universidade Federal de Sao Paulo - UNIFESP; Reumatologia, São Paulo, São Paulo
  - Centro Paulista de Investigacao Clinica - CEPIC, São Paulo, São Paulo

RESULTS

PARTICIPANT FLOW:
Groups:
- Tocilizumab: Participants received tocilizumab 8 milligrams per kilogram (mg/kg) intravenous (IV) every 4 weeks for up to 104 weeks.
Period: Overall Study
Arm/Group | Tocilizumab
Started | 23
Treated | 21
Completed | 19
Not Completed | 4
Not completed — Withdrawal by Subject | 1
Not completed — Death | 1
Not completed — Not treated | 2

BASELINE CHARACTERISTICS:
Population: Intent to treat (ITT) population included all participants who received at least 1 dose of study drug.
Groups:
- Tocilizumab: Participants received tocilizumab 8 mg/kg IV every 4 weeks for up to 104 weeks.
Arm/Group | Tocilizumab
Number analyzed (Participants) | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.5 (9.18)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 6

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Treatment Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Description: An adverse event (AE) is any unfavorable or unintended sign (including an abnormal laboratory finding), symptom or disease temporarily associated with use of study drug, regardless of its relation to study drug. A TEAE is an AE that occurs only once treatment has started. An SAE can be a) fatal, b) life-threatening, c) requires/prolongs hospitalization, d) results in persistent/significant incapacity/disability, e) results in congenital anomaly/birth defect or f) is considered as a significant medical event by the investigator.
Time Frame: Baseline up to approximately 104 weeks
Population: ITT population
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 21
percentage of participants
  TEAEs | 95.2
  SAEs | 9.5

2. Primary Outcome: Percentage of Participants With TEAEs of Special Interest
Description: An AE is any unfavorable or unintended sign (including an abnormal laboratory finding), symptom or disease temporarily associated with use of study drug, regardless of its relation to study drug. A TEAE is an AE that occurs only once treatment has started. Nine categories of AE of special interest are identified for tocilizumab which includes a) serious/medically significant infections, b) myocardial infarction/acute coronary syndrome, c) gastrointestinal perforations, d) malignancies, e) anaphylaxis/hypersensitivity reactions, f) demyelinating disorders, g) stroke, h) serious and/or medically significant bleeding events, and i) serious/medically significant hepatic events. Data reported is an average of the nine categories.
Time Frame: Baseline up to approximately 104 weeks
Population: ITT population
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 21
percentage of participants | 95.2

3. Primary Outcome: Percentage of Participants With TEAEs Leading to Change in Dose or Study Drug Discontinuation
Description: An AE is any unfavorable or unintended sign (including an abnormal laboratory finding), symptom or disease temporarily associated with use of study drug, regardless of its relation to study drug. A TEAE is an AE that occurs only once treatment has started.
Time Frame: Baseline up to approximately 104 weeks
Population: ITT population
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 21
percentage of participants
  TEAEs leading to study drug discontinuation | 4.8
  TEAEs leading to dose modification | 28.6

4. Secondary Outcome: Change From Baseline (CFB) in Disease Activity Score 28 Using Erythrocyte Sedimentation Rate (DAS28-ESR) at Specified Time Points
Description: The DAS28-ESR is a combined index for measuring disease activity in rheumatoid arthritis (RA). The index includes swollen joint counts (SJC) and tender joint counts (TJC), both scored 0-28 (higher scores indicate higher disease activity), as well as acute phase response (APR) determined as erythrocyte sedimentation rate (ESR) in millimeters per hour (mm/hr), and general health (GH) (patient global assessment of disease activity [PGA] using visual analog scale [VAS], range 1-100 millimeters [mm]) (higher scores indicate higher disease activity). DAS28-ESR is calculated according to the following formula: DAS28-ESR equals (=) [0.56 multiplied by (*) the square root (√) of TJC] plus (+) [0.28 * √ of SJC] + (0.70 * the natural logarithm [ln] ESR in mm/h) + (0.014*GH in mm VAS). DAS28-ESR scale is transformed and ranges from 0 to 10. A negative CFB indicated improvement.
Time Frame: Baseline, Weeks 12, 24, 36, 48, 56, 68, 80, 92, 104, early withdrawal (up to 104 weeks), follow-up 1 (8 weeks after the last visit or discontinuation; 112 weeks), follow-up 2 (16 weeks after the last visit or discontinuation; 120 weeks)
Population: ITT population. Here, 'n' represents the number of participants available for assessment at a given time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tocilizumab
Number analyzed (Participants) | 21
units on a scale
  Baseline (n=21) | 2.4 (1.76)
  CFB at Week 12 (n=19): number analyzed (Participants) | 19
  CFB at Week 12 (n=19) | -0.6 (1.6)
  CFB at Week 24 (n=21) | -0.6 (1.7)
  CFB at Week 36 (n=19): number analyzed (Participants) | 19
  CFB at Week 36 (n=19) | -0.5 (1.3)
  CFB at Week 48 (n=20): number analyzed (Participants) | 20
  CFB at Week 48 (n=20) | -0.6 (1.9)
  CFB at Week 56 (n=19): number analyzed (Participants) | 19
  CFB at Week 56 (n=19) | -0.5 (1.7)
  CFB at Week 68 (n=20): number analyzed (Participants) | 20
  CFB at Week 68 (n=20) | -0.4 (2.0)
  CFB at Week 80 (n=21) | 0.3 (1.9)
  CFB at Week 92 (n=18): number analyzed (Participants) | 18
  CFB at Week 92 (n=18) | -0.2 (1.5)
  CFB at Week 104 (n=16): number analyzed (Participants) | 16
  CFB at Week 104 (n=16) | -0.7 (1.3)
  CFB at Early withdrawal (n=1): number analyzed (Participants) | 1
  CFB at Early withdrawal (n=1) | -0.3 (NA) — Standard deviation (SD) is not applicable for a single participant.
  CFB at Follow-up visit 1 (n=16): number analyzed (Participants) | 16
  CFB at Follow-up visit 1 (n=16) | 0.6 (2.1)
  CFB at Follow-up visit 2 (n=14): number analyzed (Participants) | 14
  CFB at Follow-up visit 2 (n=14) | 1.7 (2.0)
Statistical Analysis 1: Comparison: Tocilizumab; Statistical analysis at Week 12; Test type: Superiority or Other; p = 0.101, Paired t-test
Statistical Analysis 2: Comparison: Tocilizumab; Statistical analysis at Week 24; Test type: Superiority or Other; p = 0.139, Paired t-test
Statistical Analysis 3: Comparison: Tocilizumab; Statistical analysis at Week 36; Test type: Superiority or Other; p = 0.116, Paired t-test
Statistical Analysis 4: Comparison: Tocilizumab; Statistical analysis at Week 48; Test type: Superiority or Other; p = 0.167, Paired t-test
Statistical Analysis 5: Comparison: Tocilizumab; Statistical analysis at Week 56; Test type: Superiority or Other; p = 0.210, Paired t-test
Statistical Analysis 6: Comparison: Tocilizumab; Statistical analysis at Week 68; Test type: Superiority or Other; p = 0.343, Paired t-test
Statistical Analysis 7: Comparison: Tocilizumab; Statistical analysis at Week 80; Test type: Superiority or Other; p = 0.533, Paired t-test
Statistical Analysis 8: Comparison: Tocilizumab; Statistical analysis at Week 92; Test type: Superiority or Other; p = 0.593, Paired t-test
Statistical Analysis 9: Comparison: Tocilizumab; Statistical analysis at Week 104; Test type: Superiority or Other; p = 0.044, Paired t-test
Statistical Analysis 10: Comparison: Tocilizumab; Statistical analysis at Follow-up visit 1; Test type: Superiority or Other; p = 0.243, Paired t-test
Statistical Analysis 11: Comparison: Tocilizumab; Statistical analysis at Follow-up visit 2; Test type: Superiority or Other; p = 0.009, Paired t-test

5. Secondary Outcome: CFB in Simplified Disease Activity Index (SDAI) Score at Specified Time Points
Description: The SDAI is a combined index for measuring disease activity. SDAI is the sum of TJC and SJC, both scored 0-28 (higher scores indicate higher disease activity), physician global assessment (PhGA) and PGA of disease activity, both scored 0 to 10 centimeters (cm) as assessed by VAS, and C-reactive protein level (CRP) in milligrams per deciliter (mg/dL) where normal is less than (<) 1 mg/dL. SDAI is calculated according to the following formula: SDAI = TJC + SJC + PhGA + PGA + CRP. SDAI ranges from 0 to 86. A negative CFB indicated improvement.
Time Frame: as for outcome 4
Population: ITT population. Here, 'n' represents the number of participants available for assessment at a given time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tocilizumab
Number analyzed (Participants) | 21
units on a scale
  Baseline (n=21) | 9.5 (11.84)
  CFB at Week 12 (n=20): number analyzed (Participants) | 20
  CFB at Week 12 (n=20) | -2.4 (7.75)
  CFB at Week 24 (n=21) | -2.7 (11.46)
  CFB at Week 36 (n=20): number analyzed (Participants) | 20
  CFB at Week 36 (n=20) | -2.8 (9.85)
  CFB at Week 48 (n=20): number analyzed (Participants) | 20
  CFB at Week 48 (n=20) | -3.0 (12.71)
  CFB at Week 56 (n=20): number analyzed (Participants) | 20
  CFB at Week 56 (n=20) | -3.2 (11.09)
  CFB at Week 68 (n=20): number analyzed (Participants) | 20
  CFB at Week 68 (n=20) | -0.6 (18.1)
  CFB at Week 80 (n=21) | 0.9 (13.92)
  CFB at Week 92 (n=19): number analyzed (Participants) | 19
  CFB at Week 92 (n=19) | -1.1 (9.47)
  CFB at Week 104 (n=19): number analyzed (Participants) | 19
  CFB at Week 104 (n=19) | -1.4 (7.6)
  CFB at Early withdrawal (n=1): number analyzed (Participants) | 1
  CFB at Early withdrawal (n=1) | -0.3 (NA) — SD is not applicable for a single participant.
  CFB at Follow-up visit 1 (n=19): number analyzed (Participants) | 19
  CFB at Follow-up visit 1 (n=19) | 2.0 (12.36)
  CFB at Follow-up visit 2 (n=14): number analyzed (Participants) | 14
  CFB at Follow-up visit 2 (n=14) | 9.5 (16.71)
Statistical Analysis 1: Comparison: Tocilizumab; Statistical analysis at Week 12; Test type: Superiority or Other; p = 0.1853, Paired t-test
Statistical Analysis 2: Comparison: Tocilizumab; Statistical analysis at Week 24; Test type: Superiority or Other; p = 0.2992, Paired t-test
Statistical Analysis 3: Comparison: Tocilizumab; Statistical analysis at Week 36; Test type: Superiority or Other; p = 0.2249, Paired t-test
Statistical Analysis 4: Comparison: Tocilizumab; Statistical analysis at Week 48; Test type: Superiority or Other; p = 0.3102, Paired t-test
Statistical Analysis 5: Comparison: Tocilizumab; Statistical analysis at Week 56; Test type: Superiority or Other; p = 0.2164, Paired t-test
Statistical Analysis 6: Comparison: Tocilizumab; Statistical analysis at Week 68; Test type: Superiority or Other; p = 0.8822, Paired t-test
Statistical Analysis 7: Comparison: Tocilizumab; Statistical analysis at Week 80; Test type: Superiority or Other; p = 0.7649, Paired t-test
Statistical Analysis 8: Comparison: Tocilizumab; Statistical analysis at Week 92; Test type: Superiority or Other; p = 0.6050, Paired t-test
Statistical Analysis 9: Comparison: Tocilizumab; Statistical analysis at Week 104; Test type: Superiority or Other; p = 0.4478, Paired t-test
Statistical Analysis 10: Comparison: Tocilizumab; Statistical analysis at Follow-up visit 1; Test type: Superiority or Other; p = 0.4821, Paired t-test
Statistical Analysis 11: Comparison: Tocilizumab; Statistical analysis at Follow-up visit 2; Test type: Superiority or Other; p = 0.0522, Paired t-test

6. Secondary Outcome: CFB in Swollen Joint Count (SJC) at Specified Time Points
Description: For SJC, a total of 66 joints are assessed. The presence of a swollen joint is scored as 1 and absence as 0. Total score is calculated by adding the scores, which ranges from 0 (best possible score or no swollen joint) to 66 (worse possible score or all swollen joints). Lower scores indicated no swollen joint and higher scores indicated worsening swollen joints.
Time Frame: Baseline, Weeks 12, 24, 36, 48, 56, 68, 80, 92, 104, follow-up 1 (8 weeks after the last visit or discontinuation; 112 weeks), follow-up 2 (16 weeks after the last visit or discontinuation; 120 weeks)
Population: ITT population. Here, 'n' represents the number of participants available for assessment at a given time point.
Measure: Mean (Standard Deviation); unit: swollen joints
Arm/Group | Tocilizumab
Number analyzed (Participants) | 21
swollen joints
  Baseline (n=21) | 0.8 (1.7)
  CFB at Week 12 (n=6): number analyzed (Participants) | 6
  CFB at Week 12 (n=6) | -1.3 (1.37)
  CFB at Week 24 (n=7): number analyzed (Participants) | 7
  CFB at Week 24 (n=7) | -1.6 (1.81)
  CFB at Week 36 (n=6): number analyzed (Participants) | 6
  CFB at Week 36 (n=6) | -1.5 (2.81)
  CFB at Week 48 (n=7): number analyzed (Participants) | 7
  CFB at Week 48 (n=7) | -0.9 (3.48)
  CFB at Week 56 (n=6): number analyzed (Participants) | 6
  CFB at Week 56 (n=6) | -1.8 (2.56)
  CFB at Week 68 (n=7): number analyzed (Participants) | 7
  CFB at Week 68 (n=7) | -2.0 (2.38)
  CFB at Week 80 (n=7): number analyzed (Participants) | 7
  CFB at Week 80 (n=7) | 1.1 (5.49)
  CFB at Week 92 (n=6): number analyzed (Participants) | 6
  CFB at Week 92 (n=6) | 1.7 (5.32)
  CFB at Week 104 (n=6): number analyzed (Participants) | 6
  CFB at Week 104 (n=6) | 1.2 (3.82)
  CFB at Follow-up visit 1 (n=6): number analyzed (Participants) | 6
  CFB at Follow-up visit 1 (n=6) | -1.3 (1.37)
  CFB at Follow-up visit 2 (n=3): number analyzed (Participants) | 3
  CFB at Follow-up visit 2 (n=3) | -1.0 (0.0)
Statistical Analysis 1: Comparison: Tocilizumab; Statistical analysis at Week 12; Test type: Superiority or Other; p = 0.0624, Paired t-test
Statistical Analysis 2: Comparison: Tocilizumab; Statistical analysis at Week 24; Test type: Superiority or Other; p = 0.0616, Paired t-test
Statistical Analysis 3: Comparison: Tocilizumab; Statistical analysis at Week 36; Test type: Superiority or Other; p = 0.2480, Paired t-test
Statistical Analysis 4: Comparison: Tocilizumab; Statistical analysis at Week 48; Test type: Superiority or Other; p = 0.5393, Paired t-test
Statistical Analysis 5: Comparison: Tocilizumab; Statistical analysis at Week 56; Test type: Superiority or Other; p = 0.1401, Paired t-test
Statistical Analysis 6: Comparison: Tocilizumab; Statistical analysis at Week 68; Test type: Superiority or Other; p = 0.0679, Paired t-test
Statistical Analysis 7: Comparison: Tocilizumab; Statistical analysis at Week 80; Test type: Superiority or Other; p = 0.6017, Paired t-test
Statistical Analysis 8: Comparison: Tocilizumab; Statistical analysis at Week 92; Test type: Superiority or Other; p = 0.4772, Paired t-test
Statistical Analysis 9: Comparison: Tocilizumab; Statistical analysis at Week 104; Test type: Superiority or Other; p = 0.4877, Paired t-test
Statistical Analysis 10: Comparison: Tocilizumab; Statistical analysis at Follow-up visit 1; Test type: Superiority or Other; p = 0.0624, Paired t-test
Statistical Analysis 11: Comparison: Tocilizumab; Statistical analysis at Follow-up visit 2; Test type: Superiority or Other; p < 0.0001, Paired t-test

7. Secondary Outcome: CFB in Tender Joint Count (TJC) at Specified Time Points
Description: The number of tender joints is recorded on the joint assessment form, no tenderness = 0, tenderness = 1, for 68 joints and joints were classified as tender/not tender giving a total possible tender joint count score of 0 to 68.
Time Frame: as for outcome 4
Population: ITT population. Here, 'n' represents the number of participants available for assessment at a given time point.
Measure: Mean (Standard Deviation); unit: tender joints
Arm/Group | Tocilizumab
Number analyzed (Participants) | 21
tender joints
  Baseline (n=21) | 5.8 (8.57)
  CFB at Week 12 (n=13): number analyzed (Participants) | 13
  CFB at Week 12 (n=13) | -3.1 (8.95)
  CFB at Week 24 (n=14): number analyzed (Participants) | 14
  CFB at Week 24 (n=14) | -4.8 (10.39)
  CFB at Week 36 (n=14): number analyzed (Participants) | 14
  CFB at Week 36 (n=14) | -5.4 (8.35)
  CFB at Week 48 (n=14): number analyzed (Participants) | 14
  CFB at Week 48 (n=14) | -5.9 (8.4)
  CFB at Week 56 (n=14): number analyzed (Participants) | 14
  CFB at Week 56 (n=14) | -6.0 (8.41)
  CFB at Week 68 (n=13): number analyzed (Participants) | 13
  CFB at Week 68 (n=13) | -2.3 (16.51)
  CFB at Week 80 (n=14): number analyzed (Participants) | 14
  CFB at Week 80 (n=14) | -3.5 (11.65)
  CFB at Week 92 (n=12): number analyzed (Participants) | 12
  CFB at Week 92 (n=12) | -3.6 (12.42)
  CFB at Week 104 (n=12): number analyzed (Participants) | 12
  CFB at Week 104 (n=12) | -4.3 (9.98)
  CFB at Early withdrawal (n=1): number analyzed (Participants) | 1
  CFB at Early withdrawal (n=1) | 0.0 (NA) — Standard deviation (SD) is not applicable for a single participant.
  CFB at Follow-up visit 1 (n=12): number analyzed (Participants) | 12
  CFB at Follow-up visit 1 (n=12) | 0.0 (0.0)
  CFB at Follow-up visit 2 (n=9): number analyzed (Participants) | 9
  CFB at Follow-up visit 2 (n=9) | 2.4 (8.85)
Statistical Analysis 1: Comparison: Tocilizumab; Statistical analysis at Week 12; Test type: Superiority or Other; p = 0.2388, Paired t-test
Statistical Analysis 2: Comparison: Tocilizumab; Statistical analysis at Week 24; Test type: Superiority or Other; p = 0.1084, Paired t-test
Statistical Analysis 3: Comparison: Tocilizumab; Statistical analysis at Week 36; Test type: Superiority or Other; p = 0.0321, Paired t-test
Statistical Analysis 4: Comparison: Tocilizumab; Statistical analysis at Week 48; Test type: Superiority or Other; p = 0.0203, Paired t-test
Statistical Analysis 5: Comparison: Tocilizumab; Statistical analysis at Week 56; Test type: Superiority or Other; p = 0.0193, Paired t-test
Statistical Analysis 6: Comparison: Tocilizumab; Statistical analysis at Week 68; Test type: Superiority or Other; p = 0.6235, Paired t-test
Statistical Analysis 7: Comparison: Tocilizumab; Statistical analysis at Week 80; Test type: Superiority or Other; p = 0.2814, Paired t-test
Statistical Analysis 8: Comparison: Tocilizumab; Statistical analysis at Week 92; Test type: Superiority or Other; p = 0.3391, Paired t-test
Statistical Analysis 9: Comparison: Tocilizumab; Statistical analysis at Week 104; Test type: Superiority or Other; p = 0.1605, Paired t-test
Statistical Analysis 10: Comparison: Tocilizumab; Statistical analysis at Follow-up visit 2; Test type: Superiority or Other; p = 0.4312, Paired t-test

8. Secondary Outcome: Percentage of Participants Reaching Clinical Remission (DAS28-ESR Score Less Than [<] 2.6 and/or SDAI Score Less Than or Equal to [</=] 3.3) Among Participants for Whom Tocilizumab Treatment Was Discontinued
Description: Remission: DAS28-ESR score <2.6 and SDAI score </=3.3. DAS28-ESR index included SJC and TJC, both scored 0-28, as well as APR determined as ESR in mm/hr, and GH (ranges 1-100 mm; higher scores=higher disease activity). DAS28=(0.56*√TJC)+(0.28*√SJC) +(0.70*ln ESR) +(0.014*GH). DAS28-ESR scale is transformed and ranges from 0 to 10. Negative CFB indicated improvement. DAS28 >2.6 (clinical remission); DAS28 2.6 to 3.2 (low disease activity); DAS28 >3.2 to 5.1 = moderate to high disease activity. SDAI is sum of TJC and SJC (both scored 0-28), PhGA and PGA of disease activity (both scored 0 to 10 cm as assessed by VAS, higher scores=higher disease activity), and CRP in mg/dL where normal is <1 mg/dL. SDAI=TJC + SJC + PhGA + PGA + CRP. SDAI ranged from 0 to 86. A negative CFB indicated improvement. SDAI <=3.3 (clinical remission), >3.4 to 11 (low disease activity) >11 to 26 (moderate disease activity), and >26 = (high/severe disease activity).
Time Frame: Baseline up to approximately 104 weeks
Population: ITT population
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 21
percentage of participants
  Percentage of participants achieved DAS28-ESR <2.6 | 100
  Percentage of participants achieved SDAI</=3.3 | 100

9. Secondary Outcome: Time to RA Crisis Among Participants Who Discontinued After Clinical Remission
Description: RA crisis is any worsening of participant disease acitivity that, in the opinion of the investigator, required intensified treatment other than supportive therapy, and may have included restart of the treatment with the study drug. Time to RA crisis is defined as the period of remission without drug until the RA crisis documentation.
Time Frame: Baseline up to approximately 104 weeks
Population: ITT population
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Tocilizumab
Number analyzed (Participants) | 21
days | 135.3 (53.73)

10. Secondary Outcome: CFB in PGA of Disease Activity Using VAS Score at Specified Time Points
Description: PGA of disease activity is assessed on a 0 to 100 mm horizontal VAS by the participant. The left-hand extreme of the line equals 0 mm, and is described as "no disease activity" (symptom-free and no arthritis symptoms) and the right-hand extreme equals 100 mm, as "maximum disease activity" (maximum arthritis disease activity). A negative CFB indicated improvement.
Time Frame: as for outcome 4
Population: ITT population. Here, 'n' represents the number of participants available for assessment at a given time point.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Tocilizumab
Number analyzed (Participants) | 21
mm
  Baseline (n=21) | 26.5 (19.90)
  CFB at Week 12 (n=20): number analyzed (Participants) | 20
  CFB at Week 12 (n=20) | -0.3 (16.1)
  CFB at Week 24 (n=21) | 2.5 (23.2)
  CFB at Week 36 (n=20): number analyzed (Participants) | 20
  CFB at Week 36 (n=20) | 2.0 (18.5)
  CFB at Week 48 (n=20): number analyzed (Participants) | 20
  CFB at Week 48 (n=20) | 0.4 (25.8)
  CFB at Week 56 (n=20): number analyzed (Participants) | 20
  CFB at Week 56 (n=20) | -0.5 (22.1)
  CFB at Week 68 (n=20): number analyzed (Participants) | 20
  CFB at Week 68 (n=20) | 1.3 (27.0)
  CFB at Week 80 (n=21) | 6.2 (27.5)
  CFB at Week 92 (n=19): number analyzed (Participants) | 19
  CFB at Week 92 (n=19) | 3.5 (21.6)
  CFB at Week 104 (n=19): number analyzed (Participants) | 19
  CFB at Week 104 (n=19) | 5.1 (18.4)
  CFB at Early withdrawal (n=1): number analyzed (Participants) | 1
  CFB at Early withdrawal (n=1) | 6.0 (NA) — SD is not applicable for a single participant.
  CFB at Follow-up visit 1 (n=17): number analyzed (Participants) | 17
  CFB at Follow-up visit 1 (n=17) | 4.9 (22.3)
  CFB at Follow-up visit 2 (n=14): number analyzed (Participants) | 14
  CFB at Follow-up visit 2 (n=14) | 11.0 (29.4)
Statistical Analysis 1: Comparison: Tocilizumab; Statistical analysis at Week 12; Test type: Superiority or Other; p = 0.934, Paired t-test
Statistical Analysis 2: Comparison: Tocilizumab; Statistical analysis at Week 24; Test type: Superiority or Other; p = 0.624, Paired t-test
Statistical Analysis 3: Comparison: Tocilizumab; Statistical analysis at Week 36; Test type: Superiority or Other; p = 0.642, Paired t-test
Statistical Analysis 4: Comparison: Tocilizumab; Statistical analysis at Week 48; Test type: Superiority or Other; p = 0.952, Paired t-test
Statistical Analysis 5: Comparison: Tocilizumab; Statistical analysis at Week 56; Test type: Superiority or Other; p = 0.928, Paired t-test
Statistical Analysis 6: Comparison: Tocilizumab; Statistical analysis at Week 68; Test type: Superiority or Other; p = 0.832, Paired t-test
Statistical Analysis 7: Comparison: Tocilizumab; Statistical analysis at Week 80; Test type: Superiority or Other; p = 0.315, Paired t-test
Statistical Analysis 8: Comparison: Tocilizumab; Statistical analysis at Week 92; Test type: Superiority or Other; p = 0.485, Paired t-test
Statistical Analysis 9: Comparison: Tocilizumab; Statistical analysis at Week 104; Test type: Superiority or Other; p = 0.246, Paired t-test
Statistical Analysis 10: Comparison: Tocilizumab; Statistical analysis at Follow-up visit 1; Test type: Superiority or Other; p = 0.375, Paired t-test
Statistical Analysis 11: Comparison: Tocilizumab; Statistical analysis at Follow-up visit 2; Test type: Superiority or Other; p = 0.185, Paired t-test

11. Secondary Outcome: CFB in PGA of Pain Using VAS Score at Specified Time Points
Description: PGA of pain is assessed on a 0 to 100 mm horizontal VAS. The left-hand extreme of the line equals 0 mm, and is described as "no pain" and the right-hand extreme equals 100 mm, and is described as "unbearable pain". A negative change indicated improvement.
Time Frame: as for outcome 4
Population: ITT population. Here, 'n' represents the number of participants available for assessment at a given time point.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Tocilizumab
Number analyzed (Participants) | 21
mm
  Baseline (n=21) | 22.3 (21.76)
  CFB at Week 12 (n=20): number analyzed (Participants) | 20
  CFB at Week 12 (n=20) | 2.5 (14.1)
  CFB at Week 24 (n=21) | 5.0 (27.7)
  CFB at Week 36 (n=20): number analyzed (Participants) | 20
  CFB at Week 36 (n=20) | 3.6 (18.5)
  CFB at Week 48 (n=20): number analyzed (Participants) | 20
  CFB at Week 48 (n=20) | 0.6 (26.4)
  CFB at Week 56 (n=20): number analyzed (Participants) | 20
  CFB at Week 56 (n=20) | 1.0 (20.0)
  CFB at Week 68 (n=20): number analyzed (Participants) | 20
  CFB at Week 68 (n=20) | 3.7 (26.4)
  CFB at Week 80 (n=21) | 7.5 (28.9)
  CFB at Week 92 (n=19): number analyzed (Participants) | 19
  CFB at Week 92 (n=19) | 2.8 (23.4)
  CFB at Week 104 (n=19): number analyzed (Participants) | 19
  CFB at Week 104 (n=19) | 5.8 (19.8)
  CFB at Early withdrawal (n=1): number analyzed (Participants) | 1
  CFB at Early withdrawal (n=1) | 8.0 (NA) — SD is not applicable for a single participant.
  CFB at Follow-up visit 1 (n=17): number analyzed (Participants) | 17
  CFB at Follow-up visit 1 (n=17) | 7.8 (24.4)
  CFB at Follow-up visit 2 (n=14): number analyzed (Participants) | 14
  CFB at Follow-up visit 2 (n=14) | 13.6 (29.0)
Statistical Analysis 1: Comparison: Tocilizumab; Statistical analysis at Week 12; Test type: Superiority or Other; p = 0.445, Paired t-test
Statistical Analysis 2: Comparison: Tocilizumab; Statistical analysis at Week 24; Test type: Superiority or Other; p = 0.414, Paired t-test
Statistical Analysis 3: Comparison: Tocilizumab; Statistical analysis at Week 36; Test type: Superiority or Other; p = 0.401, Paired t-test
Statistical Analysis 4: Comparison: Tocilizumab; Statistical analysis at Week 48; Test type: Superiority or Other; p = 0.920, Paired t-test
Statistical Analysis 5: Comparison: Tocilizumab; Statistical analysis at Week 56; Test type: Superiority or Other; p = 0.834, Paired t-test
Statistical Analysis 6: Comparison: Tocilizumab; Statistical analysis at Week 68; Test type: Superiority or Other; p = 0.539, Paired t-test
Statistical Analysis 7: Comparison: Tocilizumab; Statistical analysis at Week 80; Test type: Superiority or Other; p = 0.246, Paired t-test
Statistical Analysis 8: Comparison: Tocilizumab; Statistical analysis at Week 92; Test type: Superiority or Other; p = 0.602, Paired t-test
Statistical Analysis 9: Comparison: Tocilizumab; Statistical analysis at Week 104; Test type: Superiority or Other; p = 0.218, Paired t-test
Statistical Analysis 10: Comparison: Tocilizumab; Statistical analysis at Follow-up visit 1; Test type: Superiority or Other; p = 0.208, Paired t-test
Statistical Analysis 11: Comparison: Tocilizumab; Statistical analysis at Follow-up visit 2; Test type: Superiority or Other; p = 0.101, Paired t-test

12. Secondary Outcome: CFB in PhGA of Disease Activity Using VAS Score at Specified Time Points
Description: PhGA of disease activity is assessed on a 0 to 100 mm horizontal VAS by the physician. The left-hand extreme of the line equals 0 mm, and is described as "no disease activity" (symptom-free and no arthritis symptoms) and the right-hand extreme equals 100 mm as "maximum disease activity" (maximum arthritis disease activity).
Time Frame: as for outcome 4
Population: ITT population. Here, 'n' represents the number of participants available for assessment at a given time point.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Tocilizumab
Number analyzed (Participants) | 21
mm
  Baseline (n=21) | 7.9 (11.13)
  CFB at Week 12 (n=20): number analyzed (Participants) | 20
  CFB at Week 12 (n=20) | -1.0 (7.3)
  CFB at Week 24 (n=21) | -0.8 (7.7)
  CFB at Week 36 (n=20): number analyzed (Participants) | 20
  CFB at Week 36 (n=20) | -1.0 (8.3)
  CFB at Week 48 (n=20): number analyzed (Participants) | 20
  CFB at Week 48 (n=20) | 0.8 (13.1)
  CFB at Week 56 (n=20): number analyzed (Participants) | 20
  CFB at Week 56 (n=20) | -2.2 (9.6)
  CFB at Week 68 (n=20): number analyzed (Participants) | 20
  CFB at Week 68 (n=20) | 1.5 (18.1)
  CFB at Week 80 (n=21) | 7.6 (21.3)
  CFB at Week 92 (n=19): number analyzed (Participants) | 19
  CFB at Week 92 (n=19) | 4.1 (13.3)
  CFB at Week 104 (n=19): number analyzed (Participants) | 19
  CFB at Week 104 (n=19) | 5.1 (12.2)
  CFB at Early withdrawal (n=1): number analyzed (Participants) | 1
  CFB at Early withdrawal (n=1) | -1.0 (NA) — SD is not applicable for a single participant.
  CFB at Follow-up visit 1 (n=19): number analyzed (Participants) | 19
  CFB at Follow-up visit 1 (n=19) | 3.4 (9.0)
  CFB at Follow-up visit 2 (n=14): number analyzed (Participants) | 14
  CFB at Follow-up visit 2 (n=14) | 9.1 (17.3)
Statistical Analysis 1: Comparison: Tocilizumab; Statistical analysis at Week 12; Test type: Superiority or Other; p = 0.565, Paired t-test
Statistical Analysis 2: Comparison: Tocilizumab; Statistical analysis at Week 24; Test type: Superiority or Other; p = 0.637, Paired t-test
Statistical Analysis 3: Comparison: Tocilizumab; Statistical analysis at Week 36; Test type: Superiority or Other; p = 0.594, Paired t-test
Statistical Analysis 4: Comparison: Tocilizumab; Statistical analysis at Week 48; Test type: Superiority or Other; p = 0.788, Paired t-test
Statistical Analysis 5: Comparison: Tocilizumab; Statistical analysis at Week 56; Test type: Superiority or Other; p = 0.329, Paired t-test
Statistical Analysis 6: Comparison: Tocilizumab; Statistical analysis at Week 68; Test type: Superiority or Other; p = 0.716, Paired t-test
Statistical Analysis 7: Comparison: Tocilizumab; Statistical analysis at Week 80; Test type: Superiority or Other; p = 0.119, Paired t-test
Statistical Analysis 8: Comparison: Tocilizumab; Statistical analysis at Week 92; Test type: Superiority or Other; p = 0.201, Paired t-test
Statistical Analysis 9: Comparison: Tocilizumab; Statistical analysis at Week 104; Test type: Superiority or Other; p = 0.087, Paired t-test
Statistical Analysis 10: Comparison: Tocilizumab; Statistical analysis at Follow-up visit 1; Test type: Superiority or Other; p = 0.116, Paired t-test
Statistical Analysis 11: Comparison: Tocilizumab; Statistical analysis at Follow-up visit 2; Test type: Superiority or Other; p = 0.070, Paired t-test

13. Secondary Outcome: CFB in Health Assessment Questionnaire-Disease Index (HAQ-DI) Score at Specified Time Points
Description: HAQ-DI is a self-reported participant questionnaire specific for RA. It consists of 20 questions referring to 8 domains: dressing/grooming, arising, eating, walking, hygiene, reach, grip; common daily activities. Each domain has at least 2 component questions. There are 4 possible responses for each component 0=without any difficulty 1=with some difficulty 2=with much difficulty 3=unable to do. Total score for HAQ-DI is the sum of all questions and ranges from 0 = without any difficulty to 60 = unable to do. A negative CFB indicates improvement.
Time Frame: as for outcome 4
Population: ITT population. Here, 'n' represents the number of participants available for assessment at a given time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tocilizumab
Number analyzed (Participants) | 21
units on a scale
  Baseline (n=21) | 4.38 (5.463)
  CFB at Week 12 (n=20): number analyzed (Participants) | 20
  CFB at Week 12 (n=20) | 1.60 (7.155)
  CFB at Week 24 (n=21) | -0.10 (4.560)
  CFB at Week 36 (n=20): number analyzed (Participants) | 20
  CFB at Week 36 (n=20) | 0.05 (4.419)
  CFB at Week 48 (n=20): number analyzed (Participants) | 20
  CFB at Week 48 (n=20) | -1.05 (4.199)
  CFB at Week 56 (n=20): number analyzed (Participants) | 20
  CFB at Week 56 (n=20) | -0.65 (4.258)
  CFB at Week 68 (n=20): number analyzed (Participants) | 20
  CFB at Week 68 (n=20) | -0.40 (7.373)
  CFB at Week 80 (n=21) | 2.57 (10.03)
  CFB at Week 92 (n=19): number analyzed (Participants) | 19
  CFB at Week 92 (n=19) | 1.21 (5.855)
  CFB at Week 104 (n=19): number analyzed (Participants) | 19
  CFB at Week 104 (n=19) | 0.21 (5.473)
  CFB at Early withdrawal (n=1): number analyzed (Participants) | 1
  CFB at Early withdrawal (n=1) | -1.00 (NA) — SD is not applicable for a single participant.
  CFB at Follow-up visit 1 (n=17): number analyzed (Participants) | 17
  CFB at Follow-up visit 1 (n=17) | 0.94 (5.226)
  CFB at Follow-up visit 2 (n=14): number analyzed (Participants) | 14
  CFB at Follow-up visit 2 (n=14) | 3.64 (6.344)
Statistical Analysis 1: Comparison: Tocilizumab; Statistical analysis at Week 12; Test type: Superiority or Other; p = 0.3299, Paired t-test
Statistical Analysis 2: Comparison: Tocilizumab; Statistical analysis at Week 24; Test type: Superiority or Other; p = 0.9247, Paired t-test
Statistical Analysis 3: Comparison: Tocilizumab; Statistical analysis at Week 36; Test type: Superiority or Other; p = 0.9602, Paired t-test
Statistical Analysis 4: Comparison: Tocilizumab; Statistical analysis at Week 48; Test type: Superiority or Other; p = 0.2773, Paired t-test
Statistical Analysis 5: Comparison: Tocilizumab; Statistical analysis at Week 56; Test type: Superiority or Other; p = 0.5031, Paired t-test
Statistical Analysis 6: Comparison: Tocilizumab; Statistical analysis at Week 68; Test type: Superiority or Other; p = 0.8109, Paired t-test
Statistical Analysis 7: Comparison: Tocilizumab; Statistical analysis at Week 80; Test type: Superiority or Other; p = 0.2540, Paired t-test
Statistical Analysis 8: Comparison: Tocilizumab; Statistical analysis at Week 92; Test type: Superiority or Other; p = 0.3794, Paired t-test
Statistical Analysis 9: Comparison: Tocilizumab; Statistical analysis at Week 104; Test type: Superiority or Other; p = 0.8687, Paired t-test
Statistical Analysis 10: Comparison: Tocilizumab; Statistical analysis at Follow-up visit 1; Test type: Superiority or Other; p = 0.4685, Paired t-test
Statistical Analysis 11: Comparison: Tocilizumab; Statistical analysis at Follow-up visit 2; Test type: Superiority or Other; p = 0.0511, Paired t-test

ADVERSE EVENTS:
Time Frame: Baseline up to approximately 104 weeks
Description: Only TEAEs were reported.
Arm/Group | Tocilizumab
Serious Adverse Events (participants affected / at risk) | 2/21
Other Adverse Events (participants affected / at risk) | 20/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tocilizumab (N=21)
Vaginal bleeding (Reproductive system and breast disorders) | 1
Bronchopneumonia (Respiratory, thoracic and mediastinal disorders) | 1
Cardiac arrhythimia (Cardiac disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tocilizumab (N=21)
Leukopenia (Blood and lymphatic system disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 1
Dizziness (Cardiac disorders) | 1
Tachycardia (Cardiac disorders) | 1
Diabetes mellitus (Endocrine disorders) | 1
Menstruation irregular (Endocrine disorders) | 1
Ulcerative keratitis (Eye disorders) | 1
Conjunctivitis (Eye disorders) | 1
Scleritis (Eye disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 1
Impaired healing (General disorders) | 1
Drug intolerance (General disorders) | 1
Cholestasis (Hepatobiliary disorders) | 1
Hepatic steatosis (Hepatobiliary disorders) | 1
Rheumatoid arthritis (Immune system disorders) | 1
Vaginitis Bacterial (Infections and infestations) | 2
Cellulitis (Infections and infestations) | 1
Labyrinthitis (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 4
Nasopharyngitis (Infections and infestations) | 1
Viraemia (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Chest injury (Injury, poisoning and procedural complications) | 1
Transaminases Increased (Investigations) | 2
Dyslipidaemia (Metabolism and nutrition disorders) | 5
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1
Vitamin D Deficiency (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 1
Sciatica (Musculoskeletal and connective tissue disorders) | 1
Tendonitis (Musculoskeletal and connective tissue disorders) | 1
Pyogenic Granuloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Headache (Nervous system disorders) | 1
Renal cyst (Renal and urinary disorders) | 1
Urinary Tract Infection (Renal and urinary disorders) | 2
Vaginitis Bacterial (Reproductive system and breast disorders) | 1
Menorrhagia (Reproductive system and breast disorders) | 1
Acute Sinusitis (Respiratory, thoracic and mediastinal disorders) | 1
Allergic Cough (Respiratory, thoracic and mediastinal disorders) | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Upper Respiratory Tract Infection (Respiratory, thoracic and mediastinal disorders) | 9
Nasopharyngitis (Respiratory, thoracic and mediastinal disorders) | 2
Sinusitis (Respiratory, thoracic and mediastinal disorders) | 2
Tracheobronchitis (Respiratory, thoracic and mediastinal disorders) | 3
Blepharitis (Skin and subcutaneous tissue disorders) | 1
Cellulitis (Skin and subcutaneous tissue disorders) | 1
Hypertension (Vascular disorders) | 1
Mesenteric thrombosis (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.